CLINICAL TRIAL: NCT06404749
Title: Fungal Fiber for Gut Health
Acronym: FUN4GUT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The sponsor company was dissolved, resulting in insufficient funding to continue production of the investigational dietary supplement.
Sponsor: Future Biome SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: FUN4GUT01
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Mild Gastrointestinal Symptoms in Healthy Adults; Low-grade Chronic Inflammation; Stress; Gut Health; Gut Permeability; Gut Microbiome; Immune Response; Activity of Daily Living; Nutrition, Healthy
Keywords: gut microbiome; gut health; healthy women; perimenopause; pre menopause; middle aged women; fiber; gut brain axis; low grade chronic inflammation; prebiotic
MeSH Terms: interventions — Inulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: data analysts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FB01 (Experimental): fungal fiber, 150 mg/day, oral capsules, 2 weeks
  Interventions: Dietary Supplement: fungal fiber
- inulin (Active Comparator): inulin, 3 g/day, oral capsules, 2 weeks
  Interventions: Dietary Supplement: inulin

INTERVENTIONS:
Dietary Supplement: fungal fiber — fungal fiber from mycelium
  Arms: FB01
Dietary Supplement: inulin — long chain, degree of polymerization DP>23
  Arms: inulin

SUMMARY:
This study compares effects of plant based fiber vs fungi based fiber on clinical outcomes related to gut function (immunity, emotions, stress) and explores the role of gut microbiome structure and function on individual responses.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of a signed and dated informed consent form
2. Declared willingness to comply with all study procedures and availability during the study.
3. Female, >37 years, ≤48 years
4. Healthy volunteers who have experienced at least one of the following Gastrointestinal symptoms in the last week: abdominal pain, full stomach, bloating, accidental leakage of intestinal gas, loud belching, bowel movements more frequent than usual, discomfort when eating, with a GIQLI score <121
5. Fiber intake <20g/day according to R24
6. 18.5 ≤ BMI ≤ 29.9
7. Volunteers permanently living in the Buenos Aires Metropolitan Area for at least 6 months prior to the intervention.
8. Ability to take oral capsules and willingness to comply with intervention regimen of the study.
9. Agreement to comply with lifestyle considerations during the study.

Exclusion Criteria:

1. History of chronic immune, metabolic or gastrointestinal diseases.
2. History of gastrointestinal surgery.
3. Acute illness within one week prior to screening.
4. Treatment with oral or systemic antibiotics within 3 months prior to screening.
5. Hospitalization within 3 months prior to screening.
6. Consumption of laxatives or antidiarrheals, antispasmodic agents, antacids, anti-inflammatories within three days prior to screening.
7. Current intake of fiber or prebiotics as a supplement, or probiotics as a supplement.
8. Vegan, vegetarian or on a special diet.
9. Pregnancy or breastfeeding.
10. Menopause (absence of menstruation for 12 consecutive months) or postmenopause.
11. Known allergic reactions to components of the study interventions: inulin, beta-glucan, mushrooms, magnesium stearate, microcrystalline cellulose, hydroxypropylmethylcellulose.
12. Treatment with another investigational drug or other intervention in the last 6 months.
13. Receives pharmacological intervention for the treatment of a disease
14. Any disorder that, in the opinion of the investigator, could jeopardize safety of the participant.

Ages: 38 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2024-05-03 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-24 (Actual)

PRIMARY OUTCOMES:
GastroIntestinal Quality of Life Index | From enrollment to the end of treatment at 6 weeks
  GastroIntestinal Quality of Life Index (GIQLI), self assessed questionnaire, minimum score 0 (low quality), maximum score 144 (high quality)

SECONDARY OUTCOMES:
Bristol | From the enrollment to the end of treatment at 6 weeks
  Bristol scale and frequency chart. Frequency and consistence of feces, self assessed questionnaire. Range 1 to 7. Optimal value: 4. Values 1-3: different levels of constipation. Values 6-7: different levels of diarrhea
Wisconsin Upper Respiratory Symptom Survey | From enrollment to the end of treatment at 6 weeks
  Wisconsin Upper Respiratory Symptom Survey (WURSS41) scale, self assessed questionnaire, range 0 (desired) to 301 (undesired)
Positive and Negative Affect Schedule | From enrollment to the end of treatment at 6 weeks
  PANAS, self assessed questionnaire. Range from 10 (lowest) to 50 (highest) for both positive and negative scale
Work Productivity and Activity Impairment | From enrollment to the end of treatment at 6 weeks
  WPAI, self assessed questionnaire, range 0 (desired) to 100 (undesired)
basal cortisol | From enrollment to the end of treatment at 6 weeks
  basal cortisol
hs-CRP | From enrollment to the end of treatment at 6 weeks
  high sensitivity C Reactive Protein
calprotectin | From enrollment to the end of treatment at 6 weeks
  fecal
Short Chain Fatty Acids | From enrollment to the end of treatment at 6 weeks
  fecal and serum SCFA

OTHER OUTCOMES:
microbiome metagenomics | from enrollment to the end of treatment at 6 weeks
  gut microbiome taxonomy: abundance, diversity
microbiome metatranscriptomics | From enrollment to the end of treatment at 6 weeks
  expression of gut microbial genes

CONTACTS AND LOCATIONS:
Overall Officials: Javier Tartaglione, Principal Investigator
Locations (1):
- Consultorios Del Dr Jorge Eduardo Tartaglione, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Yes
a decision has not been made yet
Time Frame: a decision has not been made yet
Access Criteria: a decision has not been made yet